CLINICAL TRIAL: NCT03053440
Title: A Phase 3, Randomized, Open-Label, Multicenter Study Comparing the Efficacy and Safety of the Bruton's Tyrosine Kinase (BTK) Inhibitors BGB-3111 and Ibrutinib in Subjects With Waldenström's Macroglobulinemia (WM)
Brief Title: A Study Comparing BGB-3111 and Ibrutinib in Participants With Waldenström's Macroglobulinemia (WM)
Acronym: ASPEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-3111-302; 2016-002980-33 (EudraCT Number)
Record Dates: First submitted 2017-02-07; First posted 2017-02-15 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Waldenström's Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A : Ibrutinib (Experimental): Participants with the MYD88 mutation received Ibrutinib
  Interventions: Drug: Ibrutinib
- Arm B: Zanubrutinib (Active Comparator): Participants with the MYD88 mutation received zanubrutinib
  Interventions: Drug: BGB-3111

INTERVENTIONS:
Drug: BGB-3111 — 160 mg PO BID until progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by sponsor
  Other Names: Zanubrutinib; Brukinsa
  Arms: Arm B: Zanubrutinib
Drug: Ibrutinib — 420 mg PO QD until progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by sponsor
  Other Names: IMBRUVICA
  Arms: Arm A : Ibrutinib

SUMMARY:
This study evaluated the safety, efficacy and clinical benefit of BGB-3111 (zanubrutinib) vs ibrutinib in participants with MYD88 Mutation Waldenström's Macroglobulinemia.

DETAILED DESCRIPTION:
This open-label, randomized study compared the efficacy and safety of the Bruton's Tyrosine Kinase (BTK) inhibitors BGB-3111 and ibrutinib in participants with Waldenström's Macroglobulinemia who require therapy. Participants had baseline bone marrow samples assayed for sequencing of the MYD88 gene. 201 participants with the MYD88 mutation were enrolled and randomized to receive 160 mg BGB-3111 orally twice per day (PO BID) (treatment Arm A) or to receive 420mg ibrutinib orally once per day (PO QD) (treatment Arm B) until disease progression or unacceptable toxicity.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical and definitive histologic diagnosis of WM
* Measurable disease, requiring treatment
* Participants with no prior therapy for WM, must be considered inappropriate candidates for treatment with a standard chemoimmunotherapy regimen
* Age ≥ 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate bone marrow function
* Adequate renal and hepatic function
* Electrocardiogram/multigated acquisition scan (ECHO/MUGA) demonstrating left ventricular ejection fraction (LVEF)≥ the lower limit of institutional normal
* Participants may be enrolled who relapse after autologous stem cell transplant if they are at least 3 months after transplant, and after allogeneic transplant if they are at least 6 months post-transplant.
* Females of childbearing potential must agree to use highly effective forms of birth control throughout the course of the study and at least up to 90 days after last dose of study drug. Males must have undergone sterilization- vasectomy, or utilize a barrier method
* Life expectancy of > 4 months

Key Exclusion Criteria:

* Prior exposure to a BTK inhibitor
* Evidence of disease transformation at the time of study entry
* Corticosteroids given with antineoplastic intent within 7 days, or chemotherapy given with antineoplastic intent, targeted therapy, or radiation therapy within 3 weeks, or antibody-based therapy within 4 weeks of the start of study drug
* Major surgery within 4 weeks of study treatment
* Toxicity of ≥ Grade 2 from prior anticancer therapy
* History of other active malignancies within 2 years of study entry, with exception of (1) adequately treated in-situ carcinoma of cervix; (2) localized basal cell or squamous cell carcinoma of skin; (3) previous malignancy confined and treated locally with curative intent
* Currently active, clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, any Class 3 or 4 cardiac disease within 6 months of screening
* QTcF prolongation (defined as a QTcF > 480 msec)
* Active, clinically significant Electrocardiogram (ECG) abnormalities
* Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction
* Uncontrolled active systemic infection or recent infection requiring parenteral anti-microbial therapy
* Known human immunodeficiency virus (HIV), or active hepatitis B or hepatitis C
* Pregnant or lactating women
* Any life-threatening illness, medical condition, organ system dysfunction, need for profound anticoagulation, or bleeding disorder, which, in the investigator's opinion, could compromise the subject's safety
* Any medications which are strong or moderate cytochrome P450, family 3, subfamily A (CYP3A) inhibitors or strong CYP3A inducers

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (58):
- United States (7):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (11):
  - Paratus Clinical Research Woden, Canberra, Australian Capital Territory
  - St George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Flinders Medical Centre, Bedford PK, South Australia
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Peninsula Health Frankston, Frankston, Victoria
  - Barwon Health the Geelong Hospital, Geelong, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Czechia (3):
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- Centre Leon Berard, Lyon, France
- Germany (2):
  - Srh Kliniken Landkreis Sigmaringen, Sigmaringen
  - Universitaetsklinikum Ulm, Innere Medizin Iii, Ulm
- General Hospital of Athens Alexandra, Athens, Greece
- Italy (10):
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori Irst, Meldola
  - Niguarda Cancer Center Division of Hematology, Milan
  - Aou Maggiore Della Carita, Novara
  - Irccs Policlinico San Matteo, Universita Degli Studi Di Pavi, Pavia
  - Unita Di Ematologia, Dipartimento Di Ematologia Ed Oncologia, Ravenna
  - Fondazione Policlinico A Gemelli, Roma
  - Ao Citta Della Salute E Della Scienza Di Torino Presidio O, Torino
  - Aou Santa Maria Della Misericordia Di Udine, Udine
- Netherlands (2):
  - Amsterdam Umc Amc, Amsterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (5):
  - Uniwersytecki Szpital Kliniczny W Bialymstoku, Bialystok
  - Szpital Specjalist W Brzozowie,Podkarpacki Osrodek Onkologiczny, Brzozów
  - Szpital Uniwersytecki Nr Im Dr Jana Biziela, Bydgoszcz
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów
  - Malopolskie Centrum Medyczne Sc, Krakow
- Spain (8):
  - Hospital Universitari Germans Trias I Pujol, Badalona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario Vall Dhebron, Barcelona
  - Ico H Duran I Reynals, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Start Madrid Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitari I Politecnic La Fe, Valencia
- Karolinska Universitetssjukhuset Solna, Stockholm, Sweden
- United Kingdom (7):
  - The Royal Bournemouth and Christchurch Hospitals Nhs Foundation, Bournemouth
  - Churchill Hospital Oxford University Hospital Nhs Trust, Headington
  - St Jamess Institute of Oncology, Leeds
  - Barts Health Nhs Trust, London
  - University College Hospital, London
  - Nottingham University Hospitals Nhs Trust, Nottingham
  - Plymouth Hospitals Nhs Trust, Plymouth

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Tam CS, LeBlond V, Novotny W, Owen RG, Tedeschi A, Atwal S, Cohen A, Huang J, Buske C. A head-to-head Phase III study comparing zanubrutinib versus ibrutinib in patients with Waldenstrom macroglobulinemia. Future Oncol. 2018 Sep;14(22):2229-2237. doi: 10.2217/fon-2018-0163. Epub 2018 Jun 5. PMID 29869556
- [Derived] Garcia-Sanz R, Owen RG, Jurczak W, Dimopoulos MA, McCarthy H, Cull G, Opat SS, Castillo JJ, Kersten MJ, Wahlin BE, Grosicki S, Prathikanti R, Tian T, Allewelt H, Cohen AC, Tam CS. Outcomes after transition from ibrutinib to zanubrutinib in patients with Waldenstrom macroglobulinemia from the ASPEN study. Blood Adv. 2025 Dec 23;9(24):6538-6546. doi: 10.1182/bloodadvances.2024015596. PMID 40924923
- [Derived] Heyman BM, Opat SS, Wahlin BE, Dimopoulos MC, Castillo JJ, Tedeschi A, Tam CS, Buske C, Owen RG, Leblond V, Trotman J, Barnes G, Chan WY, Schneider J, Allewelt H, Cohen A, Matous JV. Peripheral neuropathy in the phase 3 ASPEN study of Bruton tyrosine kinase inhibitors for Waldenstrom macroglobulinemia. Blood Adv. 2025 Feb 25;9(4):722-728. doi: 10.1182/bloodadvances.2024014115. PMID 39626287
- [Derived] Tedeschi A, Tam CS, Owen RG, Buske C, Leblond V, Dimopoulos M, Garcia-Sanz R, Castillo JJ, Trotman J, Treon SP, Yang K, Tang B, Allewelt H, Patel S, Chan WY, Cohen A, Chen S, Barnes G. Health-related quality of life in patients with Waldenstrom macroglobulinemia: results from the ASPEN trial. Future Oncol. 2024;20(25):1789-1798. doi: 10.1080/14796694.2024.2355079. Epub 2024 Jul 29. PMID 39072392
- [Derived] Moslehi JJ, Furman RR, Tam CS, Salem JE, Flowers CR, Cohen A, Zhang M, Zhang J, Chen L, Ma H, Brown JR. Cardiovascular events reported in patients with B-cell malignancies treated with zanubrutinib. Blood Adv. 2024 May 28;8(10):2478-2490. doi: 10.1182/bloodadvances.2023011641. PMID 38502198
- [Derived] Dimopoulos MA, Opat S, D'Sa S, Jurczak W, Lee HP, Cull G, Owen RG, Marlton P, Wahlin BE, Garcia-Sanz R, McCarthy H, Mulligan S, Tedeschi A, Castillo JJ, Czyz J, Fernandez de Larrea C, Belada D, Libby E, Matous J, Motta M, Siddiqi T, Tani M, Trneny M, Minnema MC, Buske C, Leblond V, Treon SP, Trotman J, Chan WY, Schneider J, Allewelt H, Patel S, Cohen A, Tam CS. Zanubrutinib Versus Ibrutinib in Symptomatic Waldenstrom Macroglobulinemia: Final Analysis From the Randomized Phase III ASPEN Study. J Clin Oncol. 2023 Nov 20;41(33):5099-5106. doi: 10.1200/JCO.22.02830. Epub 2023 Jul 21. PMID 37478390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 201 participants were randomized to Arm A and Arm B in 12 countries in Australia, Europe, United Kingdom and United States.
Pre-assignment Details: The screening period consisted of Days -35 to -1.
Groups:
- Arm A: Ibrutinib: Participants diagnosed with Waldenström's Macroglobulinemia (WM) with mutated MYD88 gene received 420 mg ibrutinib once daily orally until progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by sponsor
- Arm B: Zanubrutinib: Participants diagnosed with WM with mutated MYD88 gene received 160 milligrams (mg) zanubrutinib twice daily orally until progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by sponsor
Period: Overall Study
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Started | 99 | 102
Completed | 0 | 0
Not Completed | 99 | 102
Not completed — Sponsor's Decision to End the Study | 20 | 13
Not completed — Death | 18 | 14
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — Enrolled in Long-term Extension Study | 48 | 66
Not completed — Physician Decision | 2 | 1
Not completed — Participant Randomized but died before dosing | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Analysis Set: Includes all randomized participants assigned to an arm.
Groups:
- Arm A: Ibrutinib: Participants diagnosed with WM with mutated MYD88 gene received 420 mg ibrutinib once daily orally until progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by sponsor
- Arm B: Zanubrutinib: Participants diagnosed with WM with mutated MYD88 gene received 160 mg zanubrutinib twice daily orally until progressive disease, unacceptable toxicity, death, withdrawal of consent, or study termination by sponsor
- Total: Total of all reporting groups
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib | Total
Number analyzed (Participants) | 99 | 102 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.9 (8.58) | 69.2 (10.26) | 69.5 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 33 | 67
  Male | 65 | 69 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 91 | 82 | 173
  Unknown or Not Reported | 4 | 16 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 94 | 88 | 182
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Either a Complete Response (CR) or Very Good Partial Response (VGPR) Using an Adaptation of the Response Criteria Updated at the Sixth International Workshop on WM as Assessed by an Independent Review Committee (IRC)
Description: Percentage of participants with CR, defined as normal serum immunoglobulin M (IgM) levels, disappearance of monoclonal protein by immunofixation, and negative cryoglobulinemia if cryoglobulinemia was positive at baseline, or VGPR, defined as ≥90% reduction in serum IgM level from baseline or normal serum IgM values.
Time Frame: Up to approximately 2 years and 7 months
Population: Intent To Treat (ITT) Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Percentage of Participants | 19.2 [12.0 to 28.3] | 28.4 [19.9 to 38.2]
Statistical Analysis 1: Comparison: Arm A: Ibrutinib vs Arm B: Zanubrutinib; Test type: Superiority; p = 0.0921, Cochran-Mantel-Haenszel; Based on Cochran-Mantel-Haenszel test stratified by the stratification factors per interactive response technology (IRT). p value is 2-sided; Risk Difference (RD) = 10.2, 95% CI 2-sided [-1.5 to 22.0]

2. Secondary Outcome: Percentage of Participants Achieving Major Response Rate (MRR) as Assessed by IRC
Description: MRR defined as the percentage of participants achieving a best response of response of CR, defined as normal serum IgM levels, disappearance of monoclonal protein by immunofixation, and negative cryoglobulinemia if cryoglobulinemia was positive at baseline, VGPR, defined as ≥90% reduction in serum IgM level from baseline or normal serum IgM values or partial response (PR) defined as ≥50% reduction of serum IgM from baseline.
Time Frame: Up to approximately 2 years and 7 months
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Percentage of Participants | 77.8 [68.3 to 85.5] | 77.5 [68.1 to 85.1]

3. Secondary Outcome: Duration of Response (DOR) as Assessed by IRC
Description: DOR defined as the time from first determination of response (CR, VGPR or PR) until first documentation of progression or death, whichever comes first. CR is defined as normal serum IgM levels, disappearance of monoclonal protein by immunofixation, and negative cryoglobulinemia if cryoglobulinemia was positive at baseline, VGPR, is defined as ≥90% reduction in serum IgM level from baseline or normal serum IgM values or partial response (PR) is defined as ≥50% reduction of serum IgM from baseline.
Time Frame: Up to approximately 2 years and 7 months
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Months | NA [8.0 to NA] — NA = Not estimable due to insufficient number of events | NA [NA to NA] — NA = Not estimable due to insufficient number of events

4. Secondary Outcome: DOR as Assessed by IRC: Event -Free Rate
Description: Estimated percentage of participants who were event-free based on Kaplan-Meier method.
Time Frame: 12 and 18 months from the date of randomization (up to approximately 2 years and 7 months)
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Percentage of Participants
  12 Months | 87.9 [77.0 to 93.8] | 94.4 [85.8 to 97.9]
  18 Months | 87.9 [77.0 to 93.8] | 85.2 [71.7 to 92.6]

5. Secondary Outcome: Percentage of Participants Achieving Either CR or VGPR in as Assessed by the Investigator
Description: Percentage of participants with CR, defined as normal serum IgM levels, disappearance of monoclonal protein by immunofixation, and negative cryoglobulinemia if cryoglobulinemia was positive at Baseline, or VGPR, defined as ≥90% reduction in serum IgM level from baseline or normal serum IgM values.
Time Frame: Up to approximately 5 years and 5 months
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Percentage of Participants | 25.3 [17.1 to 35.0] | 38.2 [28.8 to 48.4]

6. Secondary Outcome: DOR as Assessed by the Investigator
Description: DOR is defined as the time from first determination of response (CR, VGPR or PR) until first documentation of progression or death, whichever comes first
Time Frame: Up to approximately 5 years and 5 months
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Months | NA [53.5 to NA] — NA = Not estimable due to insufficient number of events | NA [NA to NA] — NA = Not estimable due to insufficient number of events

7. Secondary Outcome: DOR as Assessed by the Investigator: Event-Free Rate
Description: Estimated percentage of participants who were event-free based on Kaplan-Meier method.
Time Frame: 24,36 and 48 months from the date of randomization (up to approximately 5 years and 5 months)
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Percentage of Participants
  24 Months | 87.7 [77.8 to 93.4] | 89.7 [80.4 to 94.7]
  36 Months | 77.5 [65.9 to 85.6] | 81.1 [70.1 to 88.4]
  48 Months | 73.9 [61.6 to 82.8] | 81.1 [70.1 to 88.4]

8. Secondary Outcome: Progression Free Survival (PFS) as Assessed by the IRC
Description: PFS as assessed by the IRC, defined as time from randomization to the first documentation of progression (per modified International Workshop on Waldenström macroglobulinemia [IWWM criteria]) or death, whichever occurs first
Time Frame: Up to approximately 2 years and 7 months
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Months | NA [NA to NA] — NA = Not estimable due to insufficient number of events | NA [NA to NA] — NA = Not estimable due to insufficient number of events

9. Secondary Outcome: PFS as Assessed by IRC: Event-Free Rate
Description: Estimated percentage of participants who were event-free based on Kaplan-Meier method
Time Frame: 12 and 18 months from the date of randomization (up to approximately 2 years and 7 months)
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Percentage of Participants
  12 Months | 87.2 [78.6 to 92.5] | 89.7 [81.7 to 94.3]
  18 Months | 83.8 [74.5 to 89.9] | 85.0 [75.2 to 91.2]

10. Secondary Outcome: PFS as Assessed by the Investigator
Description: PFS as assessed by the Investigator, defined as time from randomization to the first documentation of progression (per modified IWWM criteria) or death, whichever occurs first.
Time Frame: Up to approximately 5 years and 5 months
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Months | NA [54.4 to NA] — NA = Not estimable due ot insufficient number of events | NA [NA to NA] — NA = Not estimable due ot insufficient number of events

11. Secondary Outcome: PFS as Assessed by the Investigator: Event-Free Rate
Description: Percentage of participants who were event-free based on Kaplan-Meier method.
Time Frame: 24,36 and 48 months from the date of randomization (up to approximately 5 years and 5 months)
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Percentage of Participants
  24 Months | 80.6 [70.9 to 87.3] | 88.5 [80.2 to 93.5]
  36 Months | 74.8 [64.5 to 82.5] | 78.3 [68.4 to 85.5]
  48 Months | 67.3 [56.3 to 76.1] | 78.3 [68.4 to 85.5]

12. Secondary Outcome: Percentage of Participants With Resolution of All Treatment-precipitating Symptoms
Time Frame: Up to approximately 5 years and 5 months
Population: ITT Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Percentage of Participants | 78.6 | 79.2

13. Secondary Outcome: Percentage of Participants With an Anti-Lymphoma Effect
Description: Anti-Lymphoma Effect is defined as any reduction in bone marrow involvement by lymphoplasmacytoid lymphocytes and/or size of lymphadenopathy and/or splenomegaly by CT scan, at any time during the course of study treatment.
Time Frame: Up to approximately 5 years and 5 months
Population: ITT Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 99 | 102
Percentage of Participants | 84.2 | 78.8

14. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Up to approximately 5 years and 5 months
Population: Safety Analysis Set includes all participants who received any dose of zanubrutinib or ibrutinib
Measure: Number; unit: Number of Participants
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
Number analyzed (Participants) | 98 | 101
Number of Participants
  Participants with At Least 1 TEAE | 98 | 101
  Participants with SAEs | 50 | 59

ADVERSE EVENTS:
Time Frame: up to approximately 5 years and 5 months
Description: The Safety Analysis Set included all participants who received any dose of zanubrutinib or ibrutinib. Intent To Treat analysis set included all participants that were randomized. All-Cause Mortality was assessed in Intent To Treat Analysis Set. Serious Adverse Events and Other (Not Including Serious) Adverse Events were assessed in Safety Analysis Set.
Arm/Group | Arm A: Ibrutinib | Arm B: Zanubrutinib
All-Cause Mortality (participants affected / at risk) | 19/99 | 14/102
Serious Adverse Events (participants affected / at risk) | 50/98 | 59/101
Other Adverse Events (participants affected / at risk) | 96/98 | 99/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Ibrutinib (N=98) | Arm B: Zanubrutinib (N=101)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 2 (3)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5) | 2 (2)
Atrial flutter (Cardiac disorders) | 2 (3) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 3 (3) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Anal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral blood blister (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Amyloidosis (Immune system disorders) | 1 (1) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Cellulitis (Infections and infestations) | 2 (4) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Cryptococcal fungaemia (Infections and infestations) | 0 (0) | 1 (2)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (6)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)
Neurocryptococcosis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (3) | 1 (1)
Pneumonia (Infections and infestations) | 14 (15) | 2 (4)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (1) | 0 (0)
Post-acute COVID-19 syndrome (Infections and infestations) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (2) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Interferon gamma release assay positive (Investigations) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nodular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (3) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 1 (2)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (6)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Ibrutinib (N=98) | Arm B: Zanubrutinib (N=101)
Anaemia (Blood and lymphatic system disorders) | 22 (48) | 18 (57)
Increased tendency to bruise (Blood and lymphatic system disorders) | 5 (6) | 3 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 16 (51) | 29 (87)
Thrombocytopenia (Blood and lymphatic system disorders) | 16 (47) | 15 (61)
Angina pectoris (Cardiac disorders) | 4 (4) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 18 (24) | 7 (8)
Atrial flutter (Cardiac disorders) | 4 (4) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (4) | 1 (1)
Palpitations (Cardiac disorders) | 10 (15) | 6 (8)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 6 (6)
Tinnitus (Ear and labyrinth disorders) | 3 (4) | 6 (6)
Vertigo (Ear and labyrinth disorders) | 4 (4) | 3 (3)
Cataract (Eye disorders) | 6 (7) | 3 (4)
Conjunctival haemorrhage (Eye disorders) | 6 (10) | 5 (9)
Dry eye (Eye disorders) | 3 (3) | 2 (2)
Ocular hyperaemia (Eye disorders) | 3 (3) | 1 (1)
Retinal haemorrhage (Eye disorders) | 4 (8) | 0 (0)
Vision blurred (Eye disorders) | 6 (7) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 5 (5) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 6 (9) | 4 (5)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 4 (4)
Constipation (Gastrointestinal disorders) | 12 (18) | 20 (25)
Diarrhoea (Gastrointestinal disorders) | 36 (62) | 23 (38)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 7 (7) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 3 (4) | 3 (4)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (5) | 4 (4)
Gingival bleeding (Gastrointestinal disorders) | 5 (6) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 4 (5) | 2 (2)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 5 (9) | 2 (2)
Nausea (Gastrointestinal disorders) | 15 (22) | 19 (25)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (3) | 5 (5)
Stomatitis (Gastrointestinal disorders) | 5 (7) | 4 (4)
Vomiting (Gastrointestinal disorders) | 15 (20) | 14 (27)
Asthenia (General disorders) | 6 (9) | 9 (14)
Chest pain (General disorders) | 5 (5) | 4 (4)
Chills (General disorders) | 4 (5) | 3 (3)
Drug withdrawal syndrome (General disorders) | 2 (3) | 4 (4)
Fatigue (General disorders) | 19 (25) | 26 (49)
Gait disturbance (General disorders) | 0 (0) | 4 (4)
Influenza like illness (General disorders) | 5 (7) | 6 (9)
Malaise (General disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 22 (38) | 19 (29)
Peripheral swelling (General disorders) | 12 (12) | 5 (6)
Pyrexia (General disorders) | 12 (21) | 16 (30)
Seasonal allergy (Immune system disorders) | 2 (2) | 4 (4)
Bronchitis (Infections and infestations) | 4 (4) | 4 (4)
COVID-19 (Infections and infestations) | 5 (5) | 9 (10)
Cellulitis (Infections and infestations) | 7 (18) | 6 (10)
Conjunctivitis (Infections and infestations) | 7 (7) | 2 (3)
Cystitis (Infections and infestations) | 3 (3) | 0 (0)
Ear infection (Infections and infestations) | 3 (3) | 2 (2)
Folliculitis (Infections and infestations) | 5 (6) | 2 (2)
Furuncle (Infections and infestations) | 4 (7) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (6) | 6 (7)
Herpes zoster (Infections and infestations) | 4 (4) | 5 (5)
Laryngitis (Infections and infestations) | 3 (3) | 0 (0)
Localised infection (Infections and infestations) | 11 (15) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 10 (15) | 8 (13)
Nail infection (Infections and infestations) | 6 (11) | 0 (0)
Nasopharyngitis (Infections and infestations) | 9 (10) | 14 (21)
Onychomycosis (Infections and infestations) | 5 (5) | 1 (1)
Oral herpes (Infections and infestations) | 5 (7) | 1 (1)
Paronychia (Infections and infestations) | 3 (4) | 2 (2)
Pneumonia (Infections and infestations) | 9 (9) | 3 (3)
Respiratory tract infection (Infections and infestations) | 3 (4) | 8 (10)
Rhinitis (Infections and infestations) | 7 (8) | 7 (12)
Sinusitis (Infections and infestations) | 10 (11) | 6 (9)
Skin infection (Infections and infestations) | 7 (16) | 3 (4)
Tooth infection (Infections and infestations) | 5 (9) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 31 (55) | 33 (49)
Urinary tract infection (Infections and infestations) | 17 (38) | 16 (25)
Wound infection (Infections and infestations) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 27 (59) | 19 (38)
Fall (Injury, poisoning and procedural complications) | 10 (12) | 9 (17)
Joint injury (Injury, poisoning and procedural complications) | 4 (5) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 5 (7) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 4 (5)
Skin laceration (Injury, poisoning and procedural complications) | 8 (13) | 5 (5)
Alanine aminotransferase increased (Investigations) | 3 (5) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (6) | 2 (2)
Neutrophil count decreased (Investigations) | 4 (9) | 8 (33)
Decreased appetite (Metabolism and nutrition disorders) | 4 (6) | 4 (4)
Gout (Metabolism and nutrition disorders) | 5 (6) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (10) | 3 (4)
Hyperuricaemia (Metabolism and nutrition disorders) | 9 (14) | 4 (7)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (14)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Iron deficiency (Metabolism and nutrition disorders) | 7 (7) | 7 (8)
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (50) | 24 (42)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (23) | 18 (31)
Joint swelling (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 28 (43) | 12 (15)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 7 (9)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (12) | 15 (21)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 3 (3)
Dizziness (Nervous system disorders) | 14 (16) | 15 (29)
Headache (Nervous system disorders) | 15 (20) | 17 (20)
Neuralgia (Nervous system disorders) | 3 (3) | 0 (0)
Paraesthesia (Nervous system disorders) | 8 (10) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (6) | 8 (10)
Sciatica (Nervous system disorders) | 3 (4) | 1 (1)
Syncope (Nervous system disorders) | 6 (7) | 3 (5)
Anxiety (Psychiatric disorders) | 7 (7) | 5 (5)
Depression (Psychiatric disorders) | 4 (4) | 3 (4)
Insomnia (Psychiatric disorders) | 9 (10) | 3 (4)
Acute kidney injury (Renal and urinary disorders) | 3 (4) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 13 (17) | 11 (13)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 4 (6)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (29) | 20 (36)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (11) | 17 (22)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (35) | 18 (21)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 4 (5)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 5 (6) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (12) | 2 (5)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Nail disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 10 (10) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 5 (6) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (10) | 15 (20)
Psoriasis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 6 (9) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 19 (25) | 19 (25)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (6)
Rosacea (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (9)
Skin toxicity (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Haematoma (Vascular disorders) | 9 (11) | 5 (7)
Hypertension (Vascular disorders) | 24 (46) | 16 (20)
Hypotension (Vascular disorders) | 2 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights

DOCUMENTS (2):
  • Study Protocol (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT03053440/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03053440/SAP_001.pdf